CLINICAL TRIAL: NCT06442800
Title: Online Randomized Experiment Evaluating the Perceived Effectiveness of Alcohol Warning Labels
Brief Title: Impacts of Alcohol Warning Labels: An Online Experiment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23-1218a; 1R01AA030548-01 (NIH)
Record Dates: First submitted 2024-05-30; First posted 2024-06-04 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2024-05

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alcohol Messages (Experimental): Participants will view and rate 10 messages shown on alcohol containers.
  Interventions: Behavioral: Liver Cancer; Behavioral: Throat and Mouth Cancer; Behavioral: Colorectal Cancer; Behavioral: Multiple Cancers; Behavioral: Liver Disease; Behavioral: Hypertension; Behavioral: Dementia; Behavioral: Drinking Guidelines; Behavioral: Current Warning; Behavioral: Control

INTERVENTIONS:
Behavioral: Liver Cancer — Participants will view messages about the risk of liver cancer from alcohol consumption.
Behavioral: Throat and Mouth Cancer — Participants will view messages about the risk of throat and mouth cancer from alcohol consumption.
Behavioral: Colorectal Cancer — Participants will view messages about the risk of colorectal cancer from alcohol consumption.
Behavioral: Multiple Cancers — Participants will view messages about the risk of multiple cancers from alcohol consumption.
Behavioral: Liver Disease — Participants will view messages about the risk of liver disease from alcohol consumption.
Behavioral: Hypertension — Participants will view messages about the risk of hypertension from alcohol consumption.
Behavioral: Dementia — Participants will view messages about the risk of dementia from alcohol consumption.
Behavioral: Drinking Guidelines — Participants will view messages about guidelines for alcohol consumption.
Behavioral: Current Warning — Participants will view the current warning that is required on most alcoholic beverage containers sold in the US.
Behavioral: Control — Participants will view neutral messages unrelated to the harms of alcohol consumption.

SUMMARY:
The goal of this experiment is to examine responses to alcohol warning messages about 10 different topics among US adult alcohol consumers. The main questions this experiment aims to answer are:

Which warning topics make alcohol consumers in the US want to drink less alcohol? Which warning topics remind alcohol consumers in the US of alcohol's harms? Which warning topics help alcohol consumers in the US learn something new? There will be a total of 20 alcohol messages, 2 messages for each of the 10 topics. For each topic, participants will be randomly assigned to 1 of the 2 messages so that they view a total of 10 alcohol messages. All 10 messages will be shown in random order. Participants will rate each message on how much it makes them want to drink less alcohol, reminds them that drinking can be harmful, and teaches them something new.

DETAILED DESCRIPTION:
This study aims to determine which topics in alcohol warning labels are most effective at making US adults who consume alcohol want to drink less alcohol, which topics best remind consumers of alcohol's harms, and which topics are most likely to teach consumers something new. The survey research company NORC at the University of Chicago will recruit a sample of 1,000 US adults ages 21+ who consumed alcohol at least one time per week during the past 4 weeks.

Participants will complete a within-subjects online randomized experiment in which they view and rate messages shown on alcohol containers. Participants will rate each message on perceived message effectiveness (primary outcome), reminding of alcohol's harms (secondary outcome), and learning something new (secondary outcome). These tasks will be repeated for 10 messages, each with a different topic. There will be 9 warning topics (i.e., topics about alcohol's harms) and 1 control topic (i.e., neutral topic not about alcohol's harms). In this within-subjects experiment, the survey will present the topics in random order and participants will view 1 of 2 messages for each topic.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 and older
* Reside in the United States
* Able to complete a survey in English
* Consumed alcohol at least once per week during the past 4 weeks

Exclusion Criteria:

* Under the age of 21
* Reside outside of the United States
* Unable to complete a survey in English
* Consumed alcohol less than once per week during the past 4 weeks

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1123 (Actual)
Dates: Start 2024-09-25 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marissa Hall, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Anna Grummon, PhD, Principal Investigator — Stanford University
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will post de-identified individual participant data in a public repository.
Supporting Information: SAP, Analytic Code
Time Frame: Investigators will post individual participant data upon acceptance of any manuscripts associated with the data generated in this study.
Access Criteria: Data and code will be made publicly available.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alcohol Messages
Started | 1123
Completed >/= 90% of Survey | 1087
Completed Survey in Realistic Timeframe | 1036
Completed | 1036
Not Completed | 87

BASELINE CHARACTERISTICS:
Arm/Group | Alcohol Messages
Number analyzed (Participants) | 1036
Age, Customized [Count of Participants; unit: Participants]
  21-29 years | 115
  30-44 years | 342
  45-59 years | 247
  60 years or older | 332
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Woman | 509
  Man | 524
  Non-Binary or another gender | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10
  Asian | 39
  Black or African American | 115
  Hispanic, Latino, or Spanish | 138
  Middle Eastern or North African | 2
  Native Hawaiian or other Pacific Islander | 1
  White | 681
  Another race or ethnicity | 8
  More than one race or ethnicity | 32
  Unknown/Did not report race or ethnicity | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1036

OUTCOME MEASURES:

1. Primary Outcome: Perceived Message Effectiveness
Description: The study will assess perceived message effectiveness using 1 item: "How much does this message make you want to drink less alcohol?" Response options will range from "not at all" (coded as 1) to "a great deal" (coded as 5). Higher scores indicate more perceived message effectiveness. Survey weighted means are reported to account for NORC AmeriSpeak's sampling design to enable results to be statistically representative of the US population of drinkers age >/=21 who drink alcohol.
Time Frame: Assessed during one-time 15-minute online study survey
Population: This study compares the message effectiveness of the topic message to the control message. Messages within each topic were not compared to one another.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Alcohol Messages
Number analyzed (Participants) | 1036
score on a scale
  Multiple cancers | 2.66 (0.05)
  Dementia | 2.54 (0.05)
  Colorectal cancer | 2.52 (0.05)
  Liver cancer | 2.50 (0.05)
  Throat and mouth cancer | 2.49 (0.05)
  Liver disease | 2.46 (0.05)
  Hypertension | 2.33 (0.05)
  Current warning | 2.15 (0.05)
  Guidelines | 1.93 (0.05)
  Control | 1.35 (0.04)
Statistical Analysis 1: Comparison: Alcohol Messages; Multiple cancers vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 1.31
Statistical Analysis 2: Comparison: Alcohol Messages; Dementia vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 1.19
Statistical Analysis 3: Comparison: Alcohol Messages; Colorectal cancer vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 1.17
Statistical Analysis 4: Comparison: Alcohol Messages; Liver cancer vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 1.15
Statistical Analysis 5: Comparison: Alcohol Messages; Throat and mouth cancer vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 1.14
Statistical Analysis 6: Comparison: Alcohol Messages; Liver disease vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 1.11
Statistical Analysis 7: Comparison: Alcohol Messages; Hypertension vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.98
Statistical Analysis 8: Comparison: Alcohol Messages; Current warning vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.81
Statistical Analysis 9: Comparison: Alcohol Messages; Guidelines vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.58

2. Secondary Outcome: Reminding of Alcohol's Harms
Description: The study will assess reminding of alcohol's harms using 1 item: "How much does this message remind you that drinking alcohol can be harmful?" Response options will range from not at all (1) to a great deal (5). Higher scores indicate greater reminding of alcohol's harms. Survey weighted means are reported to account for NORC AmeriSpeak's sampling design to enable results to be statistically representative of the US population of drinkers age >/=21 who drink alcohol.
Time Frame: Assessed during one-time 15-minute online study survey
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Alcohol Messages
Number analyzed (Participants) | 1036
score on a scale
  Multiple cancers | 3.15 (0.05)
  Dementia | 2.99 (0.05)
  Colorectal cancer | 2.93 (0.05)
  Liver cancer | 3.00 (0.05)
  Throat and mouth cancer | 3.06 (0.05)
  Liver disease | 2.92 (0.05)
  Hypertension | 2.84 (0.05)
  Current warning | 2.91 (0.05)
  Guidelines | 2.33 (0.05)
  Control | 1.40 (0.04)
Statistical Analysis 1: Comparison: Alcohol Messages; Multiple cancers vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 1.75
Statistical Analysis 2: Comparison: Alcohol Messages; Dementia vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 1.59
Statistical Analysis 3: Comparison: Alcohol Messages; Colorectal cancer vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 1.54
Statistical Analysis 4: Comparison: Alcohol Messages; Liver cancer vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 1.60
Statistical Analysis 5: Comparison: Alcohol Messages; Throat and mouth cancer vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 1.66
Statistical Analysis 6: Comparison: Alcohol Messages; Liver disease vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 1.52
Statistical Analysis 7: Comparison: Alcohol Messages; Hypertension vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 1.45
Statistical Analysis 8: Comparison: Alcohol Messages; Current warning vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 1.52
Statistical Analysis 9: Comparison: Alcohol Messages; Guidelines vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.93

3. Secondary Outcome: Learning Something New
Description: The study will assess learning something new with 1 item: "Did you learn something new from this message?" Response options will be yes (1) and no (0). Proportion of participants who endorsed learning something new (i.e., answered 1). Survey weighted proportions are reported to account for NORC AmeriSpeak's sampling design to enable results to be statistically representative of the US population of drinkers age >/=21 who drink alcohol.
Time Frame: Assessed during one-time 15-minute online study survey
Measure: Number; unit: proportion of positive responses
Arm/Group | Alcohol Messages
Number analyzed (Participants) | 1036
proportion of positive responses
  Multiple cancers | 0.52
  Dementia | 0.48
  Colorectal cancer | 0.54
  Liver cancer | 0.28
  Throat and mouth cancer | 0.51
  Liver disease | 0.25
  Hypertension | 0.39
  Current warning | 0.18
  Guidelines | 0.28
  Control | 0.14
Statistical Analysis 1: Comparison: Alcohol Messages; Multiple cancers vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Difference in predicted proportions = 0.38
Statistical Analysis 2: Comparison: Alcohol Messages; Dementia vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Difference in predicted proportions = 0.34
Statistical Analysis 3: Comparison: Alcohol Messages; Colorectal cancer vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Difference in predicted proportions = 0.40
Statistical Analysis 4: Comparison: Alcohol Messages; Liver cancer vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Difference in predicted proportions = 0.14
Statistical Analysis 5: Comparison: Alcohol Messages; Throat and mouth cancer vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Difference in predicted proportions = 0.37
Statistical Analysis 6: Comparison: Alcohol Messages; Liver disease vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Difference in predicted proportions = 0.11
Statistical Analysis 7: Comparison: Alcohol Messages; Hypertension vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Difference in predicted proportions = 0.25
Statistical Analysis 8: Comparison: Alcohol Messages; Current warning vs. Control; Test type: Superiority; p = 0.02, Mixed Models Analysis; Difference in predicted proportions = 0.04
Statistical Analysis 9: Comparison: Alcohol Messages; Guidelines vs. Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Difference in predicted proportions = 0.14

ADVERSE EVENTS:
Time Frame: Adverse Events were not monitored/assessed for this one-time online survey study.
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed for the study.
Arm/Group | Alcohol Messages
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT06442800/Prot_SAP_002.pdf
  • Informed Consent Form (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/00/NCT06442800/ICF_001.pdf